CLINICAL TRIAL: NCT02481921
Title: Group Medical Visits in Heart Failure for Post-Hospitalization Follow-Up
Brief Title: Group Medical Visits in Heart Failure
Acronym: MEDIC-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 14-293; NCT02454985 (obsolete NCT alias)
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2023-12-08 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
Keywords: heart failure; self-management; group intervention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either usual care group or the MEDIC-HF group in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEDIC-HF (Experimental): Group clinic or shared medical appointment of Education & Intervention in Heart Failure
  Interventions: Behavioral: Group medical visits
- Usual Care (No Intervention): Usual care in heart failure

INTERVENTIONS:
Behavioral: Group medical visits — Group clinics or shared medical appointments where a multidisciplinary team of providers with expertise in nutrition, nursing, behavior and/or medication management join to manage heart failure in addition to and in support of, the patient's regular individual clinic visits.
  Other Names: SMA
  Arms: MEDIC-HF

SUMMARY:
The primary goal of this proposal is to improve the quality of care and outcomes for patients discharged with heart failure using an innovative multidisciplinary group intervention approach. Heart failure is a complex chronic illness where comprehensive patient-centered care is difficult and resource intensive. One potential solution is to use shared medical appointments (SMA), where a group of patients with the same disease process shared the same medical or clinic appointment. This can be provided by a multi-disciplinary team of providers with expertise in nutrition, nursing, behavior and medication management join to manage heart failure. The investigators will enroll patients from Providence, Cleveland and Phoenix VA Hospitals who were within 12 weeks of discharge from a heart failure hospitalization and/or an outpatient encounter (clinic, emergent or urgent care) that required IV diuretic therapy. Patients were randomized them to receive SMA intervention or usual care. Results from this project are expected to add an innovative intervention that could improve outcomes important for both the patient and the VA: health status, hospitalizations, and mortality.

DETAILED DESCRIPTION:
The primary goal of this research project is to improve the health status and outcomes for patients treated for heart failure (HF) via a group clinic or shared medical appointment approach where education to patients, disease monitoring and medication titration occurs. Studies have found patient self-care behaviors in HF (e.g. medication/dietary non-compliance) and health system factors (e.g. care discoordination, limited access, lack of education to patients and caregivers) played an important role in patient's health status and hospitalization risk to the extent that 50% of the readmissions were judged to be possibly/probably preventable. To address patient and system factors based on the Chronic Care Model, redesign of care delivery, via SMA's, can be a good solution to provide patient with peer support, self-management education while also performing disease monitoring and medication management in a group environment. The investigators propose a randomized controlled trial to enroll patients within 12 weeks of discharge from a heart failure hospitalization and/or an outpatient encounter (clinic, emergent or urgent care) that required IV diuretic therapy, and randomized them to receive either SMA intervention either weekly or bi-weekly for 4 total sessions versus usual care for HF. The investigators will determine, at 180 days from randomization, whether HF patients who participate in HF-SMA, as compared to patients who receive usual care:

1. Experience better cardiac health status measured by Kansas City Cardiomyopathy Questionnaire and overall health status measured by EQ5D;
2. Have fewer hospitalization or death and
3. Experience improvement in a) HF Self-Care behavior, or b) plasma BNP or NT-pro-BNP levels.

The sites will be Providence VA, Cleveland VA and Phoenix VA hospitals to enroll a total of 250 patients. The study duration will be 180 days for all patients from the time of randomization. The investigators will use stratified randomization with the following variables: enrollment in other programs for HF Clinic, support group or education, <2 hospitalizations last 6 months, left ventricular ejection fraction <40% and study site. The team will consist of a nutritionist, social worker or health psychologist, a clinical pharmacist and/or nurse practitioner, without the presence of a physician (cardiologist will be available on call). The session will contain an assessment of patient needs, theme-based disease self-management education, patient-initiated disease management discussion, and break-out sessions of individualized medication case management.

ELIGIBILITY:
Inclusion Criteria:

* All subjects >18 years old,
* within 12 weeks of discharge from a heart failure hospitalization and/or an outpatient encounter (clinic, emergent or urgent care) that required IV diuretic therapy
* able to participate in a group setting and
* able to sign informed consent, will be eligible for enrollment

Exclusion Criteria:

* Unable to attend the group sessions due to either psychiatric instability (acutely suicidal, psychotic) or organic brain injury (e.g., severe dementia, encephalopathy) that precludes self-reporting on health status
* Discharged to hospice or long-term nursing home facilities (as opposed to short-term rehab), or patients with a code status of comfort-measures-only
* Recipients of heart transplant or ventricular assist devices, patients receiving intravenous inotropic infusions for heart support, women who are pregnant, and patients with end-stage liver disease or renal disease on dialysis since these conditions would preclude them from standard HF care. All women of childbearing age will have a pregnancy test before study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Hank Wu, MD, Principal Investigator — Providence VA Medical Center, Providence, RI; Sherry Ball, PhD, Principal Investigator — Cleveland VA Health Care System, Cleveland, OH
Locations (3):
- United States (3):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen LB, Parent M, Taveira TH, Dev S, Wu WC. A Description of Patient and Provider Experience and Clinical Outcomes After Heart Failure Shared Medical Appointment. J Patient Exp. 2017 Dec;4(4):169-176. doi: 10.1177/2374373517714452. Epub 2017 Jun 20. PMID 29276763
- [Background] Wu WC, Parent M, Dev S, Hearns R, Taveira TH, Cohen L, Shell-Boyd J, Jewett-Tennant J, Marshall V, Gee J, Schaub K, LaForest S, Ball S. Group medical visits after heart failure hospitalization: Study protocol for a randomized-controlled trial. Contemp Clin Trials. 2018 Aug;71:140-145. doi: 10.1016/j.cct.2018.06.015. Epub 2018 Jun 22. PMID 29940335
- [Result] Marshall V, Jewett-Tennant J, Shell-Boyd J, Stevenson L, Hearns R, Gee J, Schaub K, LaForest S, Taveira TH, Cohen L, Parent M, Dev S, Barrette A, Oliver K, Wu WC, Ball SL. Healthcare providers experiences with shared medical appointments for heart failure. PLoS One. 2022 Feb 7;17(2):e0263498. doi: 10.1371/journal.pone.0263498. eCollection 2022. PMID 35130320
- [Result] Madrigal C, Kim J, Jiang L, Lafo J, Bozzay M, Primack J, Correia S, Erqou S, Wu WC, Rudolph JL. Delirium and Functional Recovery in Patients Discharged to Skilled Nursing Facilities After Hospitalization for Heart Failure. JAMA Netw Open. 2021 Mar 1;4(3):e2037968. doi: 10.1001/jamanetworkopen.2020.37968. PMID 33724390
- [Derived] Taveira TH, Cohen LB, Laforest SK, Oliver K, Parent M, Hearns R, Ball SL, Dev S, Wu WC. Shared Medical Appointments in Heart Failure for Post Acute Care Follow-Up: A Randomized Controlled Trial. J Am Heart Assoc. 2024 Aug 6;13(15):e035282. doi: 10.1161/JAHA.124.035282. Epub 2024 Jul 31. PMID 39082405

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDIC-HF: Shared Medical Appointments in Heart Failure: or group clinics with 4-10 patients at a time provided by a multidisciplinary team of health care professionals with expertise in nutrition, social work or health psychologist, and pharmacist or nurse practitioner on alternate fashion to provide heart failure care in in addition to and in support of, the patient's regular individual clinic visits.
- Usual Care: Usual heart failure care through individual clinic visits that includes but not limited to heart failure, nutrition, cardiology, and primary care, among others, available at the hospital
Period: Overall Study
Arm/Group | MEDIC-HF | Usual Care
Started | 117 | 125
Completed | 98 | 106
Not Completed | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDIC-HF | Usual Care | Total
Number analyzed (Participants) | 117 | 125 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 37 | 66
  >=65 years | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.7) | 68.9 (9.9) | 69.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 112 | 117 | 229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 37 | 63
  White | 89 | 84 | 173
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117 | 125 | 242
Left ventricular ejection fraction (LVEF) by Echocardiogram [Count of Participants; unit: Participants] — Left Ventricular Ejection Fraction (LVEF) is measured by echocardiogram, where a higher number is better.
  Participants
    LVEF <40% | 45 | 43 | 88
    LVEEF >=40% | 72 | 82 | 154

OUTCOME MEASURES:

1. Primary Outcome: EQ Visual Analog Scale (EQVAS)
Description: A self-reported scale that reports how good or bad the respondent's health is TODAY, where higher scores mean a better health state. Minimum = 0 "worst health you can imagine"; maximum= 100 "Best health you can imagine'.
Time Frame: 180 days
Population: 8 patients in the MEDIC-HF arm and 9 patients in the Usual Care arm died prior to the final survey. Additionally, 11 patients in the MEDC-HF arm and 10 patients in the Usual Care arm were lost to follow-up or did not complete the final survey. 1 usual care patient did not complete the 6 month survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Usual Care: Usual in-person clinic visits in heart failure
Arm/Group | MEDIC-HF | Usual Care
Number analyzed (Participants) | 117 | 125
score on a scale
  Baseline | 64.6 (18.1) | 66.8 (21.7)
  6 months: number analyzed (Participants) | 98 | 105
  6 months | 73.8 (17.1) | 67.0 (18.7)

2. Primary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ), Overall Summary Score
Description: KCCQ is self reported heart failure-specific health status over the prior two weeks, where higher scores mean a perceived better health status. Score ranges from 0-100 where higher score is better.
Time Frame: 180 days
Population: 1 patient in the MEDIC-HF arm did not complete KCCQ at baseline. 8 patients in the MEDIC-HF arm and 9 patients in the Usual Care arm died prior to the final survey. Additionally, 11 patients in the MEDIC-HF arm and 10 patients in the Usual Care arm were lost to follow-up or did not complete the final survey. 1 patient in the usual care arm did not complete EQ-VAS but completed KCCQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MEDIC-HF | Usual Care
Number analyzed (Participants) | 117 | 125
score on a scale
  Baseline: number analyzed (Participants) | 116 | 125
  Baseline | 60.4 (22.7) | 58.7 (24.5)
  6 months: number analyzed (Participants) | 98 | 106
  6 months | 70.0 (21.4) | 68.4 (23.0)

ADVERSE EVENTS:
Time Frame: 6 months from time of randomization
Description: We collected hospitalizations (SAE) and Emergency room visits (AE) through monthly contact of either phone or in-person visits, in addition to chart reviews
Groups:
- MEDIC-HF: Multidisciplinary Education & Intervention Class in Heart Failure
  Group medical visits: Or shared medical appointments where a multidisciplinary team of providers with expertise in nutrition, nursing, behavior and medication management join to manage heart failure in addition to and in support of, the patient's regular physician visits.
- Usual Care: Usual heart failure care
Arm/Group | MEDIC-HF | Usual Care
All-Cause Mortality (participants affected / at risk) | 10/117 | 10/125
Serious Adverse Events (participants affected / at risk) | 57/117 | 61/125
Other Adverse Events (participants affected / at risk) | 42/117 | 55/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC-HF (N=117) | Usual Care (N=125)
Any Hospitalizations (Cardiac disorders) | 57 (97) | 61 (125) — Number of subjects that had at least 1 hospitalization during the study period.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC-HF (N=117) | Usual Care (N=125)
Any Emergency room visits (Cardiac disorders) | 42 (98) | 55 (93) — Number of subjects that had at least 1 Emergency Room visit during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02481921/Prot_SAP_000.pdf